CLINICAL TRIAL: NCT01113736
Title: Pilot Study Evaluating the Efficacy of AlloMEM in Prevention of Intraperitoneal Adhesions & Peritoneal Regeneration After Loop Ileostomy
Brief Title: Pilot Study Evaluating the Efficacy of AlloMEM After Loop Ileostomy
Acronym: AlloMem
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Proxy Biomedical Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-09-23; 09-09-23 (Other: University Hospitals Case Medical Center)
Record Dates: First submitted 2010-04-12; First posted 2010-04-30 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Ileostomy; Stenosis; Surgical Wound Dehiscence; Peritoneal; Colorectal Surgery
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Constriction, Pathologic; Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Peritoneal Membrane: AlloMEM™ (Experimental): For use as a homologous tissue where native peritoneum is absent or traumatized. By decreasing adhesions and providing a peritoneal remodeling capacity, both the time needed for ileostomy closure and the risk of enterotomy or seromyotomy would be reduced. The combination could lead to decreased complication rates and therefore decreased morbidity for the surgical patients requiring an ileostomy.
  Interventions: Biological: AlloMEM™

INTERVENTIONS:
Biological: AlloMEM™ — To investigate whether the use of HPM in a temporary loop ileostomy is beneficial to patients.
  Other Names: Human Peritoneal Membrane

SUMMARY:
The objective of this study is to investigate whether the use of Human Peritoneal Membrane (HPM) in a temporary loop ileostomy is beneficial to patients. Benefit will be defined, for purposes of this study, as a decrease in adhesions resulting in decreased operative time during ileostomy closure, with promotion of peritoneal remodeling.

DETAILED DESCRIPTION:
A loop ileostomy is a common procedure used to divert fecal matter from anastomotic sites after abdominal surgeries. Major complications from creation and subsequent closure of a temporary loop ileostomy include: stoma retraction, stoma prolapsed, stenosis, herniation, intra-abdominal abscess, anastomotic leak, wound dehiscence. Small-bowel obstruction (SBO) was the most common complication. SBO is caused by adhesions in the surgical site, with narrowing or angulation of the intestine causing obstruction. Prevention of these adhesions may reduce the frequency with which SBO is seen after this surgery. Furthermore, surgery to close the ileostomy is complicated by the presence of adhesions which make dissection of the ileostomy difficult, and increase the risk of injury of the small intestine during dissection, prolonging the operation time in an effort to minimize risk to the patient.

AlloMEM™ is human peritoneal membrane designated by the Food and Drug Administration (FDA) for use as a homologous tissue where native peritoneum is absent or traumatized. The AlloMem™ is not regulated as a device and no 510k submission has been made by the FDA. AlloMem™ is allogeneic freeze-dried, irradiated human peritoneal membrane used as a soft tissue wound covering solely regulated under 361 HCT/P because by FDA definition it is: minimally manipulated; intended for homologous use only; does not involve the combination of cell or other tissues, and does not rely on the metabolic function of cells for its primary function. Two animal studies have shown that AlloMEM™ can help prevent intra-abdominal adhesions and provides the biological framework for peritoneal remodeling. By decreasing adhesions and providing a peritoneal remodeling capacity, both the time needed for ileostomy closure and the risk of enterotomy or seromyotomy would be reduced. The combination could lead to decreased complication rates and therefore decreased morbidity for the surgical patients requiring an ileostomy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 - 85 years old at the time of ileostomy formation
* Scheduled to undergo planned diverting loop ileostomy

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients with abdominal or pelvic abscess present at time of initial surgery
* Patients with a history of pulmonary embolism or deep vein thrombosis (DVT) within 1 year of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
If there is a decrease on adhesion formation of AlloMEM™ used in formation of a temporary loop ileostomy. | Average 1 hour during formation of ileostomy
  Change in adhesion formation will be analyzed via the primary outcome of ileostomy mobilization time during ileostomy closure and the secondary outcome of an adhesion grading scale.

SECONDARY OUTCOMES:
Decrease in operative time and a promotion of peritoneal remodeling | During 3 month ileostomy closure
  The objective of this study is therefore, to investigate whether the use of HPM in a temporary loop ileostomy is beneficial to patients. Benefit will be defined, for purposes of this study, as a decrease in adhesions resulting in decreased operative time during ileostomy closure, with promotion of peritoneal remodeling

CONTACTS AND LOCATIONS:
Overall Officials: Conor P. Delaney, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Jin J, Voskerician G, Hunter SA, McGee MF, Cavazzola LT, Schomisch S, Harth K, Rosen MJ. Human peritoneal membrane controls adhesion formation and host tissue response following intra-abdominal placement in a porcine model. J Surg Res. 2009 Oct;156(2):297-304. doi: 10.1016/j.jss.2009.04.010. Epub 2009 May 13. PMID 19628227
- [Derived] Keller DS, Champagne BJ, Stein SL, Ermlich BO, Delaney CP. Pilot study evaluating the efficacy of AlloMEM for prevention of intraperitoneal adhesions and peritoneal regeneration after loop ileostomy. Surg Endosc. 2013 Oct;27(10):3891-6. doi: 10.1007/s00464-013-3004-6. Epub 2013 May 14. PMID 23670746